CLINICAL TRIAL: NCT05654974
Title: Sexual Habits in Childhood Affect Penis Size in Later Adulthood: a Cross-sectional Study
Brief Title: Sexual Habits Affect Penis Size in Adulthood
Acronym: ShiP
Status: Completed | Type: Observational
Sponsor: University Medical Center, Kazakhstan (Other)
Responsible Party: Principal Investigator, Kuat Oshakbayev, a principal investigator, University Medical Center, Kazakhstan
Other Study IDs: 0000187
Record Dates: First submitted 2022-11-28; First posted 2022-12-16 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Observational Study
Keywords: penis size; frequency of erection; masturbation; coitus; sexual abstinence; body growth
MeSH Terms: conditions — Masturbation; Coitus; Sexual Abstinence | interventions — Weights and Measures; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: measurements and questionnaire — paper-based survey administration; erect penis length and girth measurements

SUMMARY:
Purpose: to assess in Kazakh adult males erect penis sizes, and study an influence of their natural physiological events and behavioral habits during their growing ages on their penile sizes nowadays.

Study Design: An observational cross-sectional survey pilot study using a correlational design with the intention-to-treat principle.

DETAILED DESCRIPTION:
Participants. A total of 282 adult Kazakh males from the Republic of Kazakhstan and who have been visited at the urology units of three university centers in the biggest cities of the Republic of Kazakhstan (Astana, Almaty, and Karaganda) were prospectively included in the study, which took place between January 2020 and January 2021.

Measurements of the penis erect length and girth were by two doctor-urologists according to the method of Veale D et al. (2015).

Statistical analysis. Two-tailed Student's t-test, Pearson correlation and multivariate tests of the MANOVA and MANCOVA (body height as covariate) were used.

Sample size estimation. In a cross-sectional observational study in assessment of erect penis size of Kazakh adult males we supposed that the primary interest lies in assessment of erect penis sizes in the three cities (k=3). The investigators wish to be 95% sure of detecting when the mean erect penis sizes not exceed 1 mm (i.e., 1-β=0.95, and m1=1, m2=0). The standard deviation of erect penis size is likely to be 1.56 mm (i.e. SD=1.56) with a statistical power of 95% and significance level of 2.5% with the Bonferroni correction based on one-sided hypothesis testing. At the 5% Type I error rate (i.e., α=0.05), the sample size of the survey is 196.

ELIGIBILITY:
Inclusion Criteria:

* male gender aged from 23 to 35 years
* fill out the questionnaire
* BMI ≤ 29.9 kilogram per meter square
* a male who has at least one healthy native child
* no non-communicable chronic diseases.

Exclusion Criteria:

* female gender
* BMI ≥ 30.0 kilogram per meter square
* infertility
* erectile dysfunction, previous pelvic surgery, suspected hypogonadism, penile disease, or deformity
* specific treatment with androgens
* alcohol or drug abuse
* history of alcohol consumption ≥ 30 g/day within the past 5 years.

Ages: 23 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 282 adult Kazakh males from the Republic of Kazakhstan and who have been visited at the urology units of three university centers in the biggest cities of the Republic of Kazakhstan (Astana, Almaty, and Karaganda) were prospectively included in the study, which took place between January 2020 and January 2021.
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
erect penis length and girth | baseline
  centimeter

CONTACTS AND LOCATIONS:
Overall Officials: Bibazhar Dukenbayeva, Dr., Study Director — ANADETO medical center
Locations (1):
- Kuat Pernekulovich Oshakbayev, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
we will make our data available to any investigator/reviewer on their own request, so that the personal privacy of our patients cannot be compromised